CLINICAL TRIAL: NCT01647646
Title: Real Life Effectiveness in Patients With Not Optimally Controlled Asthma: Symbicort SMART, or Other ICS/LABA With as Needed SABA
Brief Title: Real Life Effectiveness in Patients With Not Optimally Controlled Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shih-Lung Cheng, Chief, Division of Pulmonary Medicine, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97083
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: asthma; SMART; fixed dose
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symbicort (Active Comparator): We will evaluate the efficacy fot Symbicort use. The usage was 2 doses bid for one year period.
  Intervention drug: Seretide fixed doses therapy
  Interventions: Drug: Seretide
- Seretide (Experimental): In non-well asthma controlled patients, experimental study with Seretide regular doses (125 2 doses bid for one year) and higher doses (250 2 doses bid) for one year
  Interventions: Drug: Seretide

INTERVENTIONS:
Drug: Seretide — Using Symbicort and Seretide for asthma control measurements Compared with efficacy and safety
  Other Names: Symbicort compared with Seretide

SUMMARY:
In real life, the investigators will be using different strategies including SMART therapy or other ICS/LABA (medium and high dose) therapy and measure the efficacy for asthma control.

DETAILED DESCRIPTION:
1. All not-well controlled asthma patients would include the study.
2. We will compare three ways of asthma control including SMART, fixed doses with regular doses and fixed doses with higher doses
3. We will evaluate the efficacy/safety for these not-well controlled patients.

ELIGIBILITY:
Inclusion Criteria:

* asthma not well control

Exclusion Criteria:

* COPD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
the percentage of asthma total and well control | one year
  F/U clinical asthma control status and percentage of Acute exacerbation

SECONDARY OUTCOMES:
percentage of asthma acute exacerbation | one year